CLINICAL TRIAL: NCT03679221
Title: The Association of Depression With "Motoric Cognitive Risk" Syndrome in the Canadian Population
Brief Title: Motoric Cognitive Risk and Depression
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2019-1501
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Depression; Geriatrics; Neurocognitive Disorders
MeSH Terms: conditions — Depression; Neurocognitive Disorders | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 45-54 years old: divided in two subgroups: individuals with and without cardio-vascular risk factors and diseases
  Interventions: Other: Data collection
- Group 54-64 years old: divided in two subgroups: individuals with and without cardio-vascular risk factors and diseases
  Interventions: Other: Data collection
- Group 65-74 years old: divided in two subgroups: individuals with and without cardio-vascular risk factors and diseases
  Interventions: Other: Data collection
- Group 75-85 years old: divided in two subgroups: individuals with and without cardio-vascular risk factors and diseases
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — telephone interview questionnaire, in-home face-to-face interview, and data from the Collection Site

SUMMARY:
The overall objective of the proposal is to examine the association between depression and the newly reported "motoric cognitive risk" (MCR) syndrome, which is a pre-dementia syndrome combining subjective cognitive complaint (i.e.; memory complaint) with objective slow gait speed, in the Canadian population, with the baseline assessment of the Canadian Longitudinal Study on Aging (CLSA).

The Canadian and global population are continuously aging. Moreover, the number of individuals affected by dementia is on the rise. One good predictor of dementia is Motoric Cognitive Risk (MCR) syndrome. MCR syndrome is a highly prevalent, newly defined syndrome that combines slow gait and subjective cognitive complaint. Depression is also highly prevalent in the older population and can affect both cognition and gait. Thus, an overlap between MCR and depression is possible. Yet few studies have examined the association between MCR and depression, thus emphasizing the importance of further investigating this association. This project encompasses determining the association of MCR syndrome with depression in the Canadian context as a step to better understand MCR syndrome in Canada.

DETAILED DESCRIPTION:
Motoric Cognitive Risk syndrome (MCR) is a new clinical syndrome associating subjective cognitive complaint and objective slow gait speed with a high prevalence calculated around 10% in population aged 60 and above. MCR syndrome predicts mild and major neurocognitive disorders. MCR syndrome does not rely on a complex and time-consuming assessment, making it applicable to the aging population. Thus, MCR syndrome seems to be a good syndrome to identify individuals at risk of mild and major neurocognitive disorders in any type of healthcare setting.

Slow gait speed and cognitive complaint are unspecific symptoms that can apply to a wide variety of morbidities (i.e., having a disease or a symptom of disease), thus causing overlap with other syndromes which may influence the predictive value of MCR syndrome. One example of the same seen in previous literature is the overlap between MCR syndrome and Mild Cognitive Impairment (MCI) which is, a pre-dementia syndrome similar to MCR syndrome. Patients diagnosed with MCR syndrome can also be diagnosed with MCI, however, this is not always the case. It has been suggested that patients cumulating both syndromes could be more at risk of mild and major neurocognitive disorders. Similarly, anxiety, depressive symptomatology and/or clinical depression (ADSCD) may be associated with slow gait speed and cognitive complaint. Prevalence of ADSCD like MCR syndrome is high and estimated around 9%, with some age dependent variation: younger adults have a higher prevalence compared to older adults. Due to the high prevalence of both MCR syndrome and ADSCD, and in conjunction that subjective cognitive complaint (for MCR syndrome definition) has previously been extracted from an item of depressive questionnaires like Center for Epidemiologic Studies Depression scale (CESD) or Geriatric Depression Scale (GDS), there is a high probability of overlap between MCR syndrome and depression. As ADSCD is not a pre-dementia stage, an overlap between ADSCD and MCR syndrome can conversely to MCI syndrome result in a decreased risk for mild and major neurocognitive disorders.

Few studies have examined the association between ADSCD and MCR syndrome and reported diverging results. They found both significant and not significant associations between MCR syndrome and ADSCD. These mixed results may be explained by the definition used for ADSCD. For instance, studies have used depressive questionnaires or antidepressant use. Moreover, this divergence could also be related to the nature of the symptomology (e.g., anxiety or mood disorders), as well as age. Thus, it is important to examine the association between ADSCD and MCR syndrome taking in consideration these parameters.

The investigator has the opportunity with the baseline assessment of a large population-based prospective and observational study in Canada, known as the Canadian Longitudinal Study on Aging (CLSA) to better understand the parameters influencing the association between ADSCD and MCR syndrome.

ELIGIBILITY:
Inclusion Criteria:

* be participant of the comprehensive CLSA

Exclusion Criteria:

* dementia,
* mobility disability,
* no information about cognitive complaint,
* no measure of walking speed

Ages: 45 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals eligible for this study will be the participants of the CLSA
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective cognitive complaint | 1 hour
  elicited from the 60-minute interview telephone questionnaire item Chronic Conditions Tracking (CTT_19 CCT_MEMPB_TRM) done in CLSA study

SECONDARY OUTCOMES:
Slow gait speed | 1 day
  defined as gait speed that is one standard deviation (SD) or more below age-and sex-appropriate mean values

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided